CLINICAL TRIAL: NCT04601870
Title: Randomized Test of Financial Incentives for Smoking Cessation Treatment Engagement Among A Healthcare System's Universal Primary Care Population
Brief Title: Financial Incentives for Smoking Cessation Treatment Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-0717; A534253 (Other: UW Madison); SMPH/MEDICINE/GEN INT MD (Other: UW Madison); Protocol Version 1/6/2021 (Other: UW Madison); 3R35CA197573-06S1 (NIH)
Record Dates: First submitted 2020-10-19; First posted 2020-10-26 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-12

CONDITIONS: Quitting Smoking
Keywords: smoking cessation; financial incentives
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Financial Incentive (Experimental): N=180 participants randomized to not be offered monetary incentive to participate in an intervention to quit smoking.
  Interventions: Other: No Financial Incentive
- Financial Incentive (100 dollars) (Experimental): N=180 randomized participants will be offered a 100 dollar incentive to participate in an intervention to quit smoking.
  Interventions: Other: Financial Incentive (100 dollars)
- Financial Incentive (50 dollars) (Experimental): N=180 randomized participants will be offered a 50 dollar incentive to participant in an intervention to quit smoking.
  Interventions: Other: Financial Incentive (50 dollars)

INTERVENTIONS:
Other: No Financial Incentive — No monetary incentive to participate in quit planning and quit counseling with a tobacco cessation specialist.
  Arms: No Financial Incentive
Other: Financial Incentive (100 dollars) — Financial incentive (100 dollars) to participate in quit planning and quit counseling with a tobacco cessation specialist.
  Arms: Financial Incentive (100 dollars)
Other: Financial Incentive (50 dollars) — Financial incentive (50 dollars) to participate in quit planning and quit counseling with a tobacco cessation specialist.
  Arms: Financial Incentive (50 dollars)

SUMMARY:
This study is being done to see if financial incentives increase the rate at which smokers engage in cessation treatment. A total of 540 participants will be enrolled by invitation from 6 primary care clinics of the participating healthcare system. Participants will be in the study for approximately 28 weeks.

DETAILED DESCRIPTION:
In this randomized controlled trial, each patient of participating Group Health Cooperative of South Central Wisconsin (GHC-SCW) primary care clinics who is listed in the Cigarette User Registry receiving standard telephone contact from their GHC-SCW Tobacco Cessation Outreach Specialist (TCOS) to discuss tobacco use treatment options will be reminded of GHC-SCW's commitment to helping them improve their health, advised to quit smoking, offered support to quit smoking, recruited, screened, consented, and randomized over the phone to one of three conditions of financial engagement incentives. Smokers unwilling to participate in the incentivized treatment program will be offered entry into the existing GHC-SCW standard smoking cessation program. Participants in the research study will also receive smoking treatment via the existing GHC-SCW standard smoking cessation program. Participants in the research study will be told that they may receive a treatment engagement incentive, with the amount consistent with their randomized incentive condition; receipt of their assigned incentive amount is dependent upon their setting a quit date and completing two smoking cessation treatment counseling contacts. The smoking cessation treatment includes medication and 3 quit smoking counseling calls scheduled to occur after the recruitment contact call, which is the standard smoking cessation program available to all GHC-SCW patients. This program entails a brief counseling call a week (typically 5-7 days) pre-quit i.e., before the patient's target quit date (TQD), approximately 5-7 days following the TQD (Week 1), and about one month following the TQD (Week 4).

Research participants will be asked to complete brief (3 to 5 minute) assessments during each standard care smoking treatment counseling call by GHC-SCW, plus 15-25 minute research study phone interviews 3- and 6-months post-TQD for study purposes. Those claiming abstinence at the 6-month post-TQD phone interview will be asked to return to their primary care clinic to complete breath, urine, and/or saliva testing to verify abstinence from combustible tobacco. This will entail providing breath samples for carbon monoxide testing and/or a urine or saliva sample for immediate cotinine testing (no samples will be stored). Participants may also be asked to collect a saliva sample at home and return it in the mail if they do not attend a biochemical verification visit.

Primary Aims:

* To determine the relations between treatment engagement financial incentive amounts offered and likelihood of patient engagement in smoking cessation treatment.

  * Primary outcome measure: Patient engagement in smoking cessation treatment (defined as setting a TQD and completing two phone counseling calls).

Exploratory Aims

* Conduct exploratory analyses on the effects of the different incentive engagement amounts on biochemically confirmed point-prevalence abstinence 6 months post-quit-date, and determine whether incentive condition affects abstinence via effects on smoking treatment engagement (i.e., whether smoking treatment engagement mediates the relations between different engagement incentive conditions and 6-month smoking abstinence).
* To determine the incremental cost-effectiveness of the different financial engagement incentive amounts with regard to total program costs vs. usual care, net monetary benefit (NMB), cost per quit, and incremental cost-effectiveness ratios (ICERs), with the last determined with regard to cost of additional smoker recruited and each additional individual who quits smoking.
* To determine the representativeness of smoking treatment reach and smoking abstinence outcomes generated by the various engagement incentive amounts with regard to different groups of smokers: e.g., those low in socio-economic status, priority populations, different racial and ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* On Cigarette User Registry at a participating clinic
* Able to speak English or Spanish

Exclusion Criteria:

* Activated healthcare power of attorney or cognitive impairment that would preclude informed consent.
* Existing target quit date approximately 30 days from date of call to TCOS
* Current billable insurance status in EHR of Medicare or non-BadgerCare Medicaid
* Prior screening for Treatment Engagement incentive enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Fiore, MD, MPH, MBA, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification. Researchers whose proposed use of the data has been approved by an independent review committee identified for this purpose, for independent verification of study outcomes, or to conduct subsequent clinical research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months after publication of primary outcomes, and ending 5 years after that date.
Access Criteria: Proposals should be directed to [PI Michael Fiore, MD at UW-CTRI (mcf@ctri.wisc.edu)]. If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Financial Incentive | Financial Incentive (100 Dollars) | Financial Incentive (50 Dollars)
Started | 38 | 30 | 30
Completed | 38 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Financial Incentive | Financial Incentive (100 Dollars) | Financial Incentive (50 Dollars) | Total
Number analyzed (Participants) | 38 | 30 | 30 | 98
Age, Categorical [Count of Participants; unit: Participants] — Participants were categorized to 18 or above.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 38 | 30 | 30 | 98
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 17 | 46
  Male | 21 | 18 | 13 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 17 | 15 | 53
  Other than White | 14 | 12 | 13 | 39
  Unknown | 3 | 1 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Set A Target Quit Date (TQD) and Complete Phone Counseling
Description: The relation between treatment engagement financial incentive amounts offered and likelihood of patient engagement in smoking cessation treatment will be assessed by the number of participants who set a TQD and complete two phone counseling calls.
Time Frame: up to 60 days from enrollment
Population: Intent-to-treat analysis to assess overall engagement in the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | No Financial Incentive | Financial Incentive (100 Dollars) | Financial Incentive (50 Dollars)
Number analyzed (Participants) | 38 | 30 | 30
Participants | 14 | 14 | 14
Statistical Analysis 1: Comparison: No Financial Incentive vs Financial Incentive (50 Dollars); Test type: Superiority; p = 0.4137, Chi-squared; Chi squared equals 0.668 with 1 degrees of freedom; Odds Ratio (OR) = 1.5, 95% CI 2-sided [.566 to 3.973] — Odds ratio for completing counseling in $50 arm vs. $0 arm
Statistical Analysis 2: Comparison: No Financial Incentive vs Financial Incentive (100 Dollars); Test type: Superiority; p = 0.4137, Chi-squared; Chi squared equals 0.668 with 1 degrees of freedom; Odds Ratio (OR) = 1.5, 95% CI 2-sided [.566 to 3.973] — Odds ratio for completing counseling in $100 arm vs. $0 arm
Statistical Analysis 3: Comparison: No Financial Incentive vs Financial Incentive (100 Dollars) vs Financial Incentive (50 Dollars); $0 vs. $50 or $100; Test type: Superiority; p = .3383, Chi-squared; Chi squared equals 0.917 with 1 degrees of freedom; Odds Ratio (OR) = 1.5, 95% CI 2-sided [.653 to 3.446] — Odds ratio for completing counseling in $50 or $100 arm vs. $0 arm

2. Other Pre Specified Outcome: 6 Month Smoking Abstinence Rates
Description: Exploratory analysis on the effects of the different incentive engagement amounts on biochemically confirmed abstinence 6-month post quit date.
Time Frame: Biochemical confirmation of abstinence occurred within 1-9 days following completion of 6-month post quit date follow-up.
Population: Intent-to-treat analysis to assess population-based cessation rate.
Measure: Count of Participants; unit: Participants
Arm/Group | No Financial Incentive | Financial Incentive (100 Dollars) | Financial Incentive (50 Dollars)
Number analyzed (Participants) | 38 | 30 | 30
Participants | 3 | 5 | 2
Statistical Analysis 1: Comparison: No Financial Incentive vs Financial Incentive (50 Dollars); Test type: Superiority; p = .2650, Chi-squared; Chi squared equals 1.243 with 1 degrees of freedom; Odds Ratio (OR) = 2.333, 95% CI 2-sided [.5100 to 10.6751] — Odds ratio for achieving confirmed abstinence at 6 months post-tqd in $50 arm vs. $0 arm
Statistical Analysis 2: Comparison: No Financial Incentive vs Financial Incentive (100 Dollars); Test type: Superiority; p = .8472, Chi-squared; Chi squared equals 0.037 with 1 degrees of freedom; Odds Ratio (OR) = .8333, 95% CI 2-sided [.1301 to 5.3369] — Odds ratio for achieving confirmed abstinence at 6 months post-tqd in $100 arm vs. $0 arm
Statistical Analysis 3: Comparison: No Financial Incentive vs Financial Incentive (100 Dollars) vs Financial Incentive (50 Dollars); $0 vs. $50 or $100; Test type: Superiority; p = .5478, Chi-squared; Chi squared equals 0.361 with 1 degrees of freedom; Odds Ratio (OR) = 1.541, 95% CI 2-sided [.3731 to 6.3640] — Odds ratio for achieving confirmed abstinence at 6 months post-tqd in $50 or $100 arms vs. $0 arm
Statistical Analysis 4: Comparison: Financial Incentive (100 Dollars) vs Financial Incentive (50 Dollars); Test type: Superiority; p = .2276, Chi-squared; Chi squared equals 1.456 with 1 degrees of freedom; Odds Ratio (OR) = .3571, 95% CI 2-sided [.06355 to 2.0070] — Odds ratio for achieving confirmed abstinence at 6 months post-tqd in $100 arm vs. $50 arm

ADVERSE EVENTS:
Time Frame: 6 Months Post-Target Quit Date (up to 7 months on study)
Description: Adverse event information was collected by subject self-report only.
Arm/Group | No Financial Incentive | Financial Incentive (100 Dollars) | Financial Incentive (50 Dollars)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/38 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT04601870/Prot_SAP_000.pdf